CLINICAL TRIAL: NCT03648736
Title: Time Course of Circulating Myocardial Biomarkers After a TASH Procedure.
Acronym: TASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 17-164
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cardiac Insufficiency
Keywords: FGF23, TASH
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HOCM patients: selected for routine TASH procedure
  Interventions: Other: blood withdrawal

INTERVENTIONS:
Other: blood withdrawal — * peripheral-venous before TASH, day 1, 2, 3, one week and one month after TASH procedure
  * central-venous during TASH

SUMMARY:
The study evaluates the released myocardial substances in blood of HOCM patients after TASH procedure (small "controlled" myocardial infarction). This helps to identify new pathomechanisms and biomarker and thus provides a better understanding of development and progress of cardiac insufficiency.

DETAILED DESCRIPTION:
All patients who receive a TASH procedure in the Medical Clinic I routinely receive routinely implementation of arterial pressure catheter for invasive blood pressure monitoring (usually Arteria radialis) as well as a central venous catheter. Directly after the procedure, the blood is taken through the central venous catheter. The operation is then terminated as planned.

The postoperative treatment is performed according to the Standard Operating Procedures (SOPs) of the Medical clinic I -regular blood sampling is performed to monitor the patient's cardiac, renal and hepatic lab values. The patient is released on the 3-5th post-operative day.

As part of a routine outpatient visit to the Medical Clinic I 1 week and 1 month after the TASH procedure, an anamnestic record as well as a blood analysis is made. One month after the TASH procedure, an echocardiographic follow-up of the HOCM is routinely performed.

Adverse events or serious adverse events are documented, assessed and reported in accordance with GCP (good clinical practice).

ELIGIBILITY:
Inclusion Criteria:

* a clinical indication for TASH procedure
* an access to blood vessels
* a person qualified for legal acts, mentally abte to follow the instructions of study stuff

Exclusion Criteria:

* patients with severe anaemia - Hb <8 mg/dL
* patients with acute infectious diseases (e.g. pneumonia)
* patients with acute myocardial ischaemia (e.g. angina pectoris or ECG alterations under strain)
* patients with acute coronary syndrome in the last three months
* patients that were hospitalized for Acute Heart Failure during the last month and had to be treated by diuretics or inotropes
* a pregnant and/or breastfeeding women
* Persons that are located by a court or administrative decision in an Institution
* Persons with a relationship of dependency to investigator
* Persons with simultaneous participation in another clinical trial
* administration of an investigational drug 30 days before start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HOCM patients selected for routine TASH procedure
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Time course of FGF23 (c-terminal) | 1 month
  from baseline to 4 weeks after TASH procedure
Time course of FGF23 (intact) | 1 month
  from baseline to 4 weeks after TASH procedure

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stöhr, Dr. med., Principal Investigator — RWTH Aachen University, Aachen University Hospital, Medical Clinic I
Locations (1):
- Aachen University Hospital; Medical Clinic I - Cardiology, Pneumology, Angiology and Internal Intensive Medicine, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
The results of the study will be published in a scientific paper. The Ethics Committee will be informed about the results of the study.

REFERENCES:
- [Background] Jessup M, Brozena S. Heart failure. N Engl J Med. 2003 May 15;348(20):2007-18. doi: 10.1056/NEJMra021498. No abstract available. PMID 12748317
- [Background] Jessup M, Brozena SC. Epilogue: support devices for end stage heart failure. Cardiol Clin. 2003 Feb;21(1):135-9. doi: 10.1016/s0733-8651(02)00139-x. PMID 12790052
- [Background] Bui AL, Horwich TB, Fonarow GC. Epidemiology and risk profile of heart failure. Nat Rev Cardiol. 2011 Jan;8(1):30-41. doi: 10.1038/nrcardio.2010.165. Epub 2010 Nov 9. PMID 21060326
- [Background] Kenchaiah S, Narula J, Vasan RS. Risk factors for heart failure. Med Clin North Am. 2004 Sep;88(5):1145-72. doi: 10.1016/j.mcna.2004.04.016. PMID 15331311
- [Result] Faul C, Amaral AP, Oskouei B, Hu MC, Sloan A, Isakova T, Gutierrez OM, Aguillon-Prada R, Lincoln J, Hare JM, Mundel P, Morales A, Scialla J, Fischer M, Soliman EZ, Chen J, Go AS, Rosas SE, Nessel L, Townsend RR, Feldman HI, St John Sutton M, Ojo A, Gadegbeku C, Di Marco GS, Reuter S, Kentrup D, Tiemann K, Brand M, Hill JA, Moe OW, Kuro-O M, Kusek JW, Keane MG, Wolf M. FGF23 induces left ventricular hypertrophy. J Clin Invest. 2011 Nov;121(11):4393-408. doi: 10.1172/JCI46122. Epub 2011 Oct 10. PMID 21985788
- [Result] Leifheit-Nestler M, Grosse Siemer R, Flasbart K, Richter B, Kirchhoff F, Ziegler WH, Klintschar M, Becker JU, Erbersdobler A, Aufricht C, Seeman T, Fischer DC, Faul C, Haffner D. Induction of cardiac FGF23/FGFR4 expression is associated with left ventricular hypertrophy in patients with chronic kidney disease. Nephrol Dial Transplant. 2016 Jul;31(7):1088-99. doi: 10.1093/ndt/gfv421. Epub 2015 Dec 17. PMID 26681731
- [Result] Mirza MA, Larsson A, Melhus H, Lind L, Larsson TE. Serum intact FGF23 associate with left ventricular mass, hypertrophy and geometry in an elderly population. Atherosclerosis. 2009 Dec;207(2):546-51. doi: 10.1016/j.atherosclerosis.2009.05.013. Epub 2009 May 21. PMID 19524924
- [Result] Andrukhova O, Slavic S, Odorfer KI, Erben RG. Experimental Myocardial Infarction Upregulates Circulating Fibroblast Growth Factor-23. J Bone Miner Res. 2015 Oct;30(10):1831-9. doi: 10.1002/jbmr.2527. Epub 2015 May 6. PMID 25858796
- [Result] Andersen IA, Huntley BK, Sandberg SS, Heublein DM, Burnett JC Jr. Elevation of circulating but not myocardial FGF23 in human acute decompensated heart failure. Nephrol Dial Transplant. 2016 May;31(5):767-72. doi: 10.1093/ndt/gfv398. Epub 2015 Dec 13. PMID 26666498